CLINICAL TRIAL: NCT06814730
Title: A Double-blind, Randomized, Placebo-controlled, Phase 1b Study to Assess the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of THN391 in Early Alzheimer's Disease Subjects
Brief Title: A Study to Assess THN391 in Subjects With Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Therini Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THN391-NEU-102; 2024-519899-72-00 (EU CTIS Number)
Record Dates: First submitted 2024-12-24; First posted 2025-02-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease, Early Onset
Keywords: Early AD; Fibrin; Fibrinogen; amyloid pathology; Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1 (Experimental): THN391 (low dosage) or Placebo, IV-infusion
  Interventions: Drug: THN391; Drug: Placebo
- Cohort 2 (Experimental): THN391 (medium dosage) or Placebo, IV-infusion
  Interventions: Drug: THN391; Drug: Placebo
- Cohort 3 (Experimental): THN391 (high dosage) or Placebo, IV infusion
  Interventions: Drug: THN391; Drug: Placebo

INTERVENTIONS:
Drug: THN391 — THN391, IV infusion, 3*Q4W (every 4 weeks)
Drug: Placebo — Placebo for comparison with THN391, IV infusion, 3*Q4W

SUMMARY:
This is a Phase 1b study to evaluate different doses of the drug and see whether a drug is safe and how it behaves in the body.

THN391 has already been assessed in healthy people without Alzheimer's disease. This is the first study of THN391 in patients with Early Alzheimer's disease. Later studies will evaluate THN391 to see if it is effective for the treatment of Alzheimer's disease.

In this study, THN391 will be compared with a placebo (a look-alike substance that contains no drug). The study duration is approximately 6 months in which the participants will visit the clinic approximately 13 times and have 2 telephone calls with the site.

Patients who fulfill all criteria to participate in the study, will receive 3 times a monthly dose of THN391 or placebo in the clinic.

Assessments that will be done at several timepoints during the study will be blood collection, physical examinations and neurological examinations, 4x an MRI-scan of the head, 2x a spinal tap and some testing of the memory and thinking skills.

DETAILED DESCRIPTION:
This is a Phase 1b, randomized, double-blind, multi-center, placebo-controlled, multiple ascending dose trial in male and female participants, aged 65 to 85 years with Early Alzheimer's disease and cSVD.

The study duration is 6-8 months: first screening to assess eligibility, then 2 months' treatment period (3 monthly doses), followed by a 4 month follow-up period.

The trial will investigate THN391 in at least 3 dose cohorts, Depending on preliminary, blinded results of the first two cohorts, the sample sizes of the following dose cohort may be increased and/or additional dose cohorts may be added.

Eligible participants will be randomized to receive either THN391 or placebo.

Three dose administrations will be provided monthly. Participants will undergo clinical and laboratory-based safety-related assessments, as well as Pharmacodynamics (PD), immunogenicity, and blood Pharmacokinetic (PK) collections at different time points.

Assessments will include 4 brain MRIs (Magnetic Resonance Imaging), 2 spinal taps, electrocardiograms (ECGs), vital signs, physical and neurological examinations, adverse event recordings, monitoring of mental health, and tests to determine the severity of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to understand the study procedures and the risks involved and provide written informed consent before the first study-related activity
* 65 to 85 years of age (inclusive at the time of informed consent).
* Diagnosis of Early Alzheimer's Disease (AD)
* Diagnosis of cerebral Small Vessel Disease (cSVD), and having at least one of the following vascular risk factors: hypertension, Type 2 diabetes mellitus, or hyperlipidemia

Exclusion criteria:

* Diagnosis of moderate or severe dementia
* Any other medical condition except for early AD (e.g. any clinically significant neurological, psychiatric or large vessel disease) that could affect interpretation of study assessments
* Use of anticoagulant, except for either clopidogrel or low dose aspirin, unless taken simultaneously

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple doses of THN391 in Early AD subjects via AEs | From enrollment to the end of the follow-up period at week 24
  Incidence of Adverse Events (AEs)
To assess the safety and tolerability of multiple doses of THN391 in Early AD subjects via SAEs | From enrollment to the end of the follow-up period at week 24
  Incidence of Serious Adverse Events (SAEs)
To assess the pharmacokinetics (PK) of multiple doses of THN391 in Early AD subjects | From the first dosing to the end of the follow-up period at week 24
  Serum and CSF concentration of THN391 using validated analytical method at specified timepoints The PK parameters will be determined or calculated using non-compartmental analysis from the serum concentration time data for THN391. A complete list of PK parameters will be provided in the statistical analysis plan (SAP).
To assess the maximum plasma concentration (Cmax) for THN391 in Early AD subjects | From the first dosing to the end of the follow-up period at week 24
  Evaluate Cmax for serum and CSF concentration of THN391 at specified time points
To assess area under the curve concentration (AUC) for THN391 in Early AD subjects | From the first dosing to the end of the follow-up period at week 24
  Evaluate AUC for serum and CSF concentration of THN391 at specified time points
To measure the half-life (t1/2) of THN391 in Early AD subjects | From the first dosing to the end of the follow-up period at week 24
  Evaluate PK in serum and CSF concentration of THN391 at specified time points

SECONDARY OUTCOMES:
To assess the immunogenicity of multiple doses of THN391 in Early AD subjects | From the first dosing to the end of the follow-up period at week 24
  Occurrence of antidrug antibodies (ADA) to THN391
To assess the effects of THN391 on coagulation in Early AD subjects via aPTT | From enrollment to the end of the follow-up period at week 24
  Changes in activated partial thromboplastin time (aPTT)
To assess the effects of THN391 on coagulation in Early AD subjects via INR | From enrollment to the end of the follow-up period at week 24
  Changes in international normalized ratio (INR)
To assess the effects of THN391 on coagulation in Early AD subjects via PT | From enrollment to the end of the follow-up period at week 24
  Changes in prothrombin time (PT)
To assess the effects of THN391 on coagulation in Early AD subjects via platelet counts | From enrollment to the end of the follow-up period at week 24
  Changes in platelet counts

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Navia, MD, PhD, Study Director — Therini Bio, Inc.
Locations (4):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, New Hampshire
  - CTC-Netherlands, Groningen
- United Kingdom (2):
  - Scottish Brain Sciences, Edinburgh
  - University College London Hospitals, London

IPD SHARING:
Plan to Share IPD: No